CLINICAL TRIAL: NCT02896621
Title: Effect of Antihypertensive Agents on Diastolic Function in Patients With Sleep Apnea: Protocol for a Randomized Controlled Trial
Brief Title: Effect of Antihypertensive Agents on Diastolic Function in Patients With Sleep Apnea
Acronym: DOSA-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 45007115.0.0000.5327; GPPG: 150274 (Other: Hospital de Clinicas de Porto Alegre)
Record Dates: First submitted 2016-07-15; First posted 2016-09-12 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Hypertension; Sleep Apnea
Keywords: Sleep Apnea; Hypertension; Chlortalidone; Diastolic function
MeSH Terms: conditions — Hypertension; Sleep Apnea Syndromes | interventions — Chlorthalidone; Amiloride; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorthalidone plus amiloride (Experimental): Chlorthalidone plus amiloride group received 25 mg of chlortalidone and amiloride, 5 mg.
  A capsule with both drugs was taken once daily in the morning for eight weeks.
  Interventions: Drug: Chlorthalidone plus amiloride
- Amlodipine (Active Comparator): Amlodipine group received 10 mg. A capsule was taken once daily in the morning for eight weeks. Capsules of amlodipine had identical presentation of that the intervention drug.
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Chlorthalidone plus amiloride — A capsule with chlorthalidone plus amiloride was taken once daily in the morning for eight weeks.
  Other Names: Chlo+Ami
  Arms: Chlorthalidone plus amiloride
Drug: Amlodipine — A capsule of amlodipine was taken once daily in the morning for eight weeks.
  Other Names: Amlo
  Arms: Amlodipine

SUMMARY:
The investigators investigated diastolic function among patients with obstructive sleep apnea (OSA) and hypertension stage I. In this randomized controlled trial, participants were randomly allocated to one of two groups: chlorthalidone associated with amiloride or amlodipine. Randomization was carried out prior to the start of the trial by an epidemiologist out of clinic and the randomization list was stratified by gender and severity of OSA. The research team and participants were blinded to the randomization list and allocation concealment was implemented. This trial aimed to detect changes in the echocardiography parameters with the drug treatment (higher in the intervention than in the placebo group). The investigators also assess change in daytime sleepiness among participants who already have been diagnosed with OSA.

DETAILED DESCRIPTION:
This is a randomized controlled trial, with participants randomly allocated to one of two groups: chlorthalidone associated with amiloride or amlodipine. Capsules were identical presentation and the research team and participants were blinded to the allocation list. The randomization list was stratified by gender and severity of OSA (AHI: 10-25 or 26-40) and in blocks in time, with size four and six units. Randomization was carried out prior to the start of the trial and it was generated by a validated software (Random Allocator). In order to ensure the confidentiality of the allocation list, it was generated by an epidemiologist who did not maintain direct contact with participants and the identification of the study drugs was done through alphanumeric code, implemented via software (RedCap).

Adherence to treatment was measured by counting returned capsules and through the Morisky questionnaire with eight questions, validated for Portuguese. Participants underwent initial clinical evaluation prior to randomization and after eight weeks of treatment for evaluation of outcomes. Demographic characteristics (age, gender, skin color), socioeconomic level (education), previous morbidity (diabetes mellitus, stroke, acute myocardial infarction, cancer, rheumatic diseases), treatments in use (anti-diabetic, anti-depressants, non-steroidal anti-inflammatory, corticosteroids, nasal vasoconstrictor, appetite suppressants, lipid-lowering drugs) and lifestyle characteristics (smoking and drinking) were collected in a standardized way. The investigators also assess anthropometric measures such as weight, height, waist, neck and hip circumference, and bioimpedance for determination of lean and fat mass. Blood pressure was measured using a validated digital oscillometric monitor, with cuff appropriate to the arm circumference, and two measurements per visit were made. In addition, ECG was performed and biochemical parameters (creatinine, blood glucose, serum potassium, uric acid, cholesterol and fractions, C-reactive protein and NT-proBNP) were determined in the laboratory of Hospital de Clinicas de Porto Alegre.

The transthoracic echocardiography is performed by the CX-50 unit (Philips, Bothell, WA - USA) with sectoral S5-1 transducer. Ambulatory monitoring of blood pressure will be measured through the Mortara AMBULO 2400 device (Mortara, Milwaukee, WI, USA) with measures 15/15 minutes during the day and 20/20 minutes at night, within 24 hours of a working day. Polysomnography will be held in type III (home with device that measures at least 4 cardiorespiratory variables) held with handset Sonmocheck (Weinmann GmbH, Hamburg, Germany), a monitor that detects the position of the patient, the presence of apneas or hypopneas, heart rate and digital oximetry.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 70 years
* Stage I hypertension (systolic BP: 140-159 or diastolic BP: 90-99 mmHg)
* No antihypertensive treatment or use of one antihypertensive drug
* Apnea / hypopnea index: 10 to 49 AH / hour

Exclusion Criteria:

* Low life expectancy
* Indication for use of calcium channel blockers or diuretics
* Allergy medications study
* Heart failure
* Myocardial infarction
* Recent stroke (last 3 months)
* Secondary hypertension
* Participation in another clinical trial (last 6 months)
* Pregnant women

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-12-07 (Actual); Primary Completion 2016-02-23 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
E/A ratio | Change at eight weeks (end of the trial)
  E/A (mitral inflow indices) echocardiography

SECONDARY OUTCOMES:
Daytime sleepiness | Change at eight weeks (end of the trial)
  Increase in quality of life sleep-related (Functional Outcomes of Sleep Questionnaire; FOSQ-10) or reduction in daytime sleepiness (Epworth Sleepiness Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra C Fuchs, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided